CLINICAL TRIAL: NCT03715634
Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Novel Subcutaneous Depot Formulation of Buprenorphine (INDV-6200) in Healthy Volunteers
Brief Title: Study of a Novel Subcutaneous Depot Formulation of Buprenorphine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: INDV-6200-101
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naltrexone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depot buprenorphine (INDV-6200) (Experimental): Period 1 subjects will receive SL buprenorphine to confirm tolerance to product Period 2 subjects will receive depot buprenorphine
  Interventions: Drug: INDV-6200; Drug: SL Buprenorphine; Drug: Nalorex
- Placebo (Placebo Comparator): Period 1 subjects will receive SL buprenorphine to confirm tolerance to product Period 2 subjects will receive volume-matched placebo
  Interventions: Drug: Placebo; Drug: SL Buprenorphine; Drug: Nalorex

INTERVENTIONS:
Drug: INDV-6200 — Subjects will be randomized in a 3:1 ratio to receive either depot buprenorphine or volume-matched placebo
  Arms: Depot buprenorphine (INDV-6200)
Drug: Placebo — Subjects will be randomized in a 3:1 ratio to receive either depot buprenorphine or volume-matched placebo
  Arms: Placebo
Drug: SL Buprenorphine — All subjects will receive SL buprenorphine as non-investigational IMP to confirm tolerability
  Other Names: Subutex
Drug: Nalorex — Both Periods will include series of nalorex administrations to antagonize potential opioid effects from buprenorphine

SUMMARY:
INDV-6200 is being developed for the treatment of opioid dependency and is expected to provide sustained buprenorphine plasma concentrations. The study will be done in healthy volunteers and will administer a non-therapeutic dose of INDV-6200. Study Period 1 will evaluate the oral tolerability of sublingual (SL) buprenorphine dosed over 3 days. Period 2 will administer the investigational medicinal product (IMP) or volume matched placebo.

DETAILED DESCRIPTION:
INDV-6200 is a novel buprenorphine subcutaneous (SC) depot formulation being developed for the treatment of opioid dependency. It is expected to provide sustained buprenorphine plasma concentrations to achieve consistent and optimal occupancy of mu-opioid receptors in the brain, for the treatment of opioid use disorder. A related subcutaneously injected, extended-release product of buprenorphine base has demonstrated sustained therapeutic plasma levels of buprenorphine over a minimum of 1 month.

Extensive experience gained from RBP-6000 allowed the development of an allometric model which has been used to predict the in vivo performance of INDV-6200. The preclinical pharmacokinetic (PK) data and the predictions from allometric scaling indicate that INDV-6200 is expected to display a similar PK profile as RBP-6000. Therefore, the main objective of this study is to investigate the PK properties of this new, related formulation using a low dose with a large safety margin.

Period 1 will be used to evaluate the oral tolerability of SL buprenorphine (SUBUTEX; non-investigational medicinal product [nIMP]) dosed over 3 days. Period 2 will involve administration of the IMP (INDV-6200) or volume-matched placebo; (low dose in Cohort A or alternative dose in optional Cohort B), to evaluate PK and safety of this novel formulation.

Both periods will also include a series of Nalorex (nIMP) administrations to antagonise potential opioid effects from buprenorphine.

Based on modeling and simulation, the dose proposed for Cohort A is expected to give similar plasma buprenorphine exposure to that obtained with the same SC dose of RBP-6000. If buprenorphine plasma exposure is lower than predicted, there is an optional second cohort (Cohort B), which may be used to explore another dose level of INDV-6200 predicted.

As this is a Phase I study, using a non-therapeutic dose of INDV-6200, the most relevant population is healthy subjects as this allows a characterisation of safety, tolerability and PK for a new molecular entity in a homogeneous population without potential biases from a patient population. In order to avoid any interaction with other medication, no co-medication will be allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating females
2. Body mass index of 18.0-33.0 kg/m2 or, if outside the range, considered not clinically significant by the Investigator
3. Willing and able to communicate and participate in the whole study
4. Provide written informed consent prior to any study specific procedures
5. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment, ECG, and laboratory investigations
6. Males and females must agree to use an adequate method of contraception
7. Tolerated SL buprenorphine and nalorex during Period 1

Exclusion Criteria:

1. Medical history of opioid-related adverse reactions
2. History of clinically significant alcohol/drug abuse in the previous 5 years
3. Received any investigational medicinal product within the previous 3 months
4. Study site employees or immediate family members of study site or sponsor employee
5. Previously enrolled in the study
6. Regular alcohol consumption in males greater than 21 units/week and females greater than 14 units/week
7. Current smokers and those who have smoked within the last 6 months
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 6 months
9. Do not have suitable veins for multiple venipunctures
10. Clinically significant abnormal biochemistry, haematology or urinalysis
11. Positive urine drug screen at screening and admission for each period
12. Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results
13. History of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory, or gastrointestinal disease, or psychiatric disorder
14. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
15. Clinically significant allergy requiring treatment. Hayfever is allowed unless active
16. Donation or loss of greater than 400 mL of blood within the previous 3 months
17. Taking or have taken, any prescribed or over-the counter drugs or herbal remedies in the 14 days before IMP administrations. Exceptions may apply
18. Injection sites containing any skin discolouration, tattoo, scar tissue or other abnormalities that may impair injection site assessment
19. Any food or drink containing grapefruit or Seville oranges within 7 days prior to first dose of buprenorphine
20. Treatment with any known drugs that are moderate or strong inhibitors/inducers of cytochrome P450 (CYP) 3A4 and/or cytochrome 450 2C8 enzyme within 30 days prior to first dose of study drug
21. Clinically significant abnormal ECG, including QT interval corrected using Fridericia's formula of greater than 450msec in males and greater than 470 msec in females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Assessment of PK of INDV-6200 (buprenorphine) | 84 days
  The key parameter of the time of maximum concentration (Tmax) of buprenorphine will be evaluated.
Assessment of PK of INDV-6200 (buprenorphine) | 84 days
  The key parameter of the maximum concentration (Cmax) of buprenorphine will be evaluated.
Assessment of PK of INDV-6200 (buprenorphine) | 84 days
  The key parameter of the cumulative area under the curve (AUC) for each PK sample will be evaluated.
Assessment of PK of INDV-6200 (buprenorphine) | 84 days
  The key parameter of the half life of buprenorphine will be evaluated.

SECONDARY OUTCOMES:
Assessment of PK of INDV-6200 (norbuprenorphine) | 84 days
  The key parameter of Tmax of norbuprenorphine will be evaluated.
Assessment of PK INDV-6200 (norbuprenorphine) | 84 days
  The key parameter of Cmax of norbuprenorphine will be evaluated.
Assessment of PK of INDV-6200 (norbuprenorphine) | 84 days
  The key parameter of the half life of norbuprenorphine will be evaluated
Assessment of PK of INDV-6200 (norbuprenorphine) | 84 days
  The key parameter of the cumulative area under the curve (AUC) for each PK sample will be evaluated.
Incidence of treatment emergence adverse events (TEAE) as assessed by changes in physical examination. | Through day 84
  Targeted physical examination will be performed focusing on abnormalities identified at screening and any changes. Clinically significant changes will be reported as adverse events (AE)
Incidence of treatment emergence adverse events (TEAE) as assessed by changes in liver function tests. | Through day 84
  Laboratory data will be summarized and any clinically significant abnormality will be reported as an AE
Incidence of treatment emergence adverse events (TEAE) as assessed by changes in systolic and diastolic blood pressure | Through day 84
  Blood pressure measurements (systolic and diastolic) will be summarized and any clinically significant abnormality will be reported as an AE
Incidence of treatment emergence adverse events (TEAE) as assessed by changes in heart rate | Through day 84
  Heart rate will be summarized and any clinically significant changes will be reported as an AE
Incidence of treatment emergence adverse events (TEAE) as assessed by electrocardiogram (ECG) changes | Through day 84
  ECG intervals will be measured and summarized and any clinically significant changes will be reported as an AE
Incidence of treatment emergence adverse events (TEAE) through assessment of the injection site for incidence of erythema | Through day 84
  Injection site assessment will be performed by the investigator using a 4 point scale. Levels of erythema will be summarized using counts and percentages at each timepoint by treatment
Incidence of treatment emergence adverse events (TEAE) through assessment of the injection site for incidence of swelling | Through day 84
  Injection site assessment will be performed by the investigator using a 4 point scale. Levels of swelling will be summarized using counts and percentages at each timepoint by treatment
Incidence of treatment emergence adverse events (TEAE) through assessment of the injection site for incidence of pain | Through day 84
  Injection site assessment will be performed by the investigator using a 4 point scale. Levels of pain will be summarized using counts and percentages at each timepoint by treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No